CLINICAL TRIAL: NCT00671983
Title: The Effect of Obstructive Sleep Apnea on Medical and Neurobehavioral Outcomes After Gastric Bypass Surgery - An Exploratory Investigation
Brief Title: The Effect of Obstructive Sleep Apnea on Medical Outcomes After Gastric Bypass Surgery
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: not adequate resources
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anthony Doufas, Principle Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SU-04282008-1124; 11812
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Sleep Apnea, Obstructive
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

INTERVENTIONS:
Procedure: Neurocognitive Testing

SUMMARY:
Obstructive sleep apnea (OSA) is a syndrome characterized by repetitive episodes of airway obstruction during sleep, which result in low oxygen level in the blood and bad sleep quality. Both of these effects are implicated in medical, neurological and cognitive disorders in subjects with OSA. The purpose of this study is to examine how OSA affects medical and neurobehavioral outcomes after gastric bypass surgery for weight loss in morbidly obese patients.

ELIGIBILITY:
Inclusion Criteria:

Scheduled for Laparoscopic roux-en-Y gastric bypass (RYGB) surgery Presence or absence of OSA confirmed by polysomnography Comprehension of spoken and written English

Exclusion Criteria:

Major psychiatric, neurological, or neuromuscular disorder History of untreated thyroid disease Known diabetes mellitus History of stroke with or without apparent neurological deficits Alcohol consumption which exceeds 2 drinks per day or drug abuse. Undergone a sleep study in the past

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
The effect of preoperative OSA on the long term neurocognitive function after Roux-en-Y gastric bypass (RYGB) surgery for weight loss in morbidly obese patients | 1 year after surgery

SECONDARY OUTCOMES:
The effect of preoperative neurocognitive impairment on the long term neurocognitive function after RYGB | 1 year after surgery
The effect of preoperative neurocognitive impairment on the weight loss function after RYGB and how this relates to the presence of OSA | 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Doufas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States